CLINICAL TRIAL: NCT06019754
Title: The One-Point Puncture Anterior Approach of the Combined Lumbar and Sacral Plexuses Block for Analgesia of Lower Limb Orthopedic Surgeries
Brief Title: Combined Lumbar and Sacral Branches Block Through the Ilio-Psoas Muscle Spaces for Analgesia of Lower Limb Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Naglaa Fathy Abdelhaleem Abdelhaleem, Lecturer, Anesthesia and Surgical Intensive Care department, Faculty of Medicine, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB#10892
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2023-08

CONDITIONS: Lower Limb Fracture
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Using a point puncture approach instead of two punctures to perform lumbosacral plexuses block in the interventional group.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Randomization assignments will be kept in sealed envelopes until all preprocedural measurements will be completed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Placebo Comparator): patients who will be recruited in the control group will receive general anesthesia only
  Interventions: Procedure: one point combined Lumbar and sacral plexus block
- Interventional group (Active Comparator): Patients who will be recruited in the Interventional will receive one point combined lumbar and sacral plexus block. then they will receive general anesthesia
  Interventions: Procedure: one point combined Lumbar and sacral plexus block

INTERVENTIONS:
Procedure: one point combined Lumbar and sacral plexus block — performing an ultrasound-guided one-point combined Lumbar and sacral plexus block using a one-point puncture. Block success will be assessed using the perfusion index (PI) before and after performing the block
  Other Names: No block intervention in control group

SUMMARY:
lumbosacral plexus block (LSPB) has been widely applied in orthopedics departments due to its advantages, including reduction in the application of opiates, decreasing the occurrence of acute pain, promoting early activation, and shortening the time of hospital stay. LSPB is a peripheral regional technique of anesthesia and analgesia, that provides a block of the main components of the lumbosacral plexus.

DETAILED DESCRIPTION:
Traditional ultrasound-guided lumbar plexus block combined with sacral plexus block requires separate blocks at different sites, requiring the lateral decubitus or prone position, which may be suboptimal in patients with severe pain. we present an anterior approach for combined lumbar and sacral plexus blocks with a one-point puncture.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II.
* patients scheduled for unilateral femur or tibial surgery necessitate knee joint intervention
* patients who have severe pain hindering changing their position or patients who have spinal fractures or refusing spinal anesthesia.
* patients with the capability of communication

Exclusion Criteria:

* puncture site infection
* patients with coagulation disorders
* patients who refuse to participate or withdraw due to personal reasons
* allergy to local anesthetics.
* past surgery at the site of the block
* hip ankylosis
* drug abuse
* Body mass index ≥ 35 kg/m2
* peripheral vascular insufficiency
* use of alpha or beta blocker agents
* Nerve injury or neuropathy of the affected lower limb
* cardiovascular or respiratory decompansation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-04 (Actual)

PRIMARY OUTCOMES:
Total intraoperative and postoperative opioid consumption | Total fentanyl used intraoperative and total morphine consumed up to 24 hours postoperative
  The total fentanyl doses consumed in the entire operative procedure and morphine consumed for 24 hours postoperative will be calculated.

SECONDARY OUTCOMES:
(NRS) score assessment pre-block, 30 min post-block , and postoperatively in the recovery room, and then it will be repeated 3 h, 6h, 12h, and 24, hours | preoperative and postoperatively pain (NRS) score assessment for 24 hours
  Numerical Pain Score (NRS) ranges from 0 to 10, where 0 is no pain, and 10 is the worst pain imaginable. Adequate pain control will be considered at Numerical Pain Score (NRS) < 4.
  Pain will be assessed using (the NRS) score preoperatively before the block and 30 min post-block, then postoperatively in the recovery room, 3 h, 6h, 12h, and 24 hours.
Block success assessment using perfusion index (PI) before and after performing the block | Recording Perfusion index readings at baseline and 10, 20, 30 min. post block
  Perfusion index (PI) values rise with successful peripheral nerve blocks. If PI is not changed, this means block failure

CONTACTS AND LOCATIONS:
Overall Officials: Naglaa Abdelhaleem, MD, Principal Investigator — Faculty of medicine, Zagazig University Hospitals
Locations (1):
- Faculty of Medicine - Zagazig University, Zagazig, Egypt